CLINICAL TRIAL: NCT00248755
Title: Pilot Study of a New Technique for Assessing Mucociliary Clearance and Airway Surface Liquid Volume in Cystic Fibrosis
Brief Title: Assessing Mucociliary Clearance and Airway Liquid Volume in the CF Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Tim Corcoran, Associate Professor of Medicine and Bioengineering, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CFFR883
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; mucociliary clearance; nuclear medicine
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Procedure: mucociliary clearance scan

SUMMARY:
The objective of this study is to determine the effect of airway surface liquid (ASL) volume on mucociliary clearance in cystic fibrosis (CF). A two-isotope nuclear medicine technique will be utilized. This pilot trial will include the imaging of n=7 CF subjects and n=7 healthy subjects. The trial will include one study visit per subject that will take approximately 3 hours. Hypothesis: The simultaneous imaging of both a "floating" and a "penetrating" radioisotope tag will allow the relative effect of airway surface liquid volume on mucociliary clearance to be determined when evaluated in CF and normal subjects.

DETAILED DESCRIPTION:
Improper function of the mucociliary clearance system in the Cystic Fibrosis (CF) lung is a major factor contributing to the chronic respiratory manifestations of the disease. Normally this host defense mechanism removes inhaled pathogens and toxins from the inner surfaces of the lung. In CF, mutations in the CF gene result in dysfunction of the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) ion channel on the cells that line the airway epithelium, causing improper fluxes of ions such as sodium, chloride, and bicarbonate. The so called "low volume" hypothesis of CF pathogenesis contends that the liquid lining the airways becomes very thin and viscous due to abnormal absorption of sodium from the airways, which draws water out of the airways, partially or totally defeating mucociliary clearance. The rate at which the mucociliary system clears materials from the lungs can be quantified using a nuclear medicine test called a mucociliary clearance scan. This study pilots a new variation of the mucociliary clearance scan that uses both "floating" and "penetrating" radioisotope tags. The difference in clearance between these tags will provide information on how airway surface liquid volume affects mucociliary clearance. This pilot trial will include the imaging of n=5 CF subjects and n=5 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of cystic fibrosis as determined by sweat test or genotype and clinical symptoms (CF subjects only)
* Clinically stable as determined by the investigator (pulmonologist)

Exclusion Criteria:

* Reactive airways disease
* Tobacco smokers
* Positive urine pregnancy test on the day of testing
* FEV1p value of < 30%
* SaO2 < 92%, or if they require supplemental oxygen.
* Subjects receiving other radioisotope treatments within the last 2 weeks will be excluded.
* Normal subjects with any history of lung disease will be excluded.
* Women currently breastfeeding an infant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14
Dates: Start 2005-11; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
radioisotope clearance rates-comparison between healthy and cf subjects

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E Corcoran, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Corcoran TE, Thomas KM, Myerburg MM, Muthukrishnan A, Weber L, Frizzell R, Pilewski JM. Absorptive clearance of DTPA as an aerosol-based biomarker in the cystic fibrosis airway. Eur Respir J. 2010 Apr;35(4):781-6. doi: 10.1183/09031936.00059009. Epub 2009 Aug 28. PMID 19717485